CLINICAL TRIAL: NCT06177262
Title: Characteristics of Illness Awareness and Its Evolution in Relation to Clinical, Cognitive and Psychosocial Variables in Anorexia Nervosa
Brief Title: Characteristics of Illness Awareness in Anorexia Nervosa
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Collaborators: Hospital Mutua de Terrassa (Other)
Responsible Party: Sponsor
Other Study IDs: IIBSP-INS-2021-122
Record Dates: First submitted 2022-11-17; First posted 2023-12-20 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-06

CONDITIONS: Insight Impaired
MeSH Terms: interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: cognitive behavioral therapy — Cognitive behavioral therapy for eating disorders.

SUMMARY:
Objective: To study the characteristics of illness awareness, its dimensions and its evolution in relation to clinical, cognitive and psychosocial variables in patients with anorexia nervosa.

Design: observational longitudinal design. Method: First, the process of translating and culturally adapting the Schedule for the Assessment of Insight in Eating Disorders (SAI-ED) to Spanish will be carried out and, over 9 months, patients who are admitted to the Eating Disorders Unit of the Hospital de la Santa Creu I Sant Pau (HSCSP) and the Eating Disorders Unit of the H. Mutua de Terrassa will be offered to participate in the study. Through individual clinical interviews and self-reports, a first sample will be collected to allow the validation study of the scale in the Spanish population.

The sample will include patients with Anorexia Nervosa and Bulimia Nervosa who understand and speak Spanish or Catalan and sign the informed consent for participation. Participants will be recruited consecutively until N=80 is reached.

From a subsample of patients with anorexia nervosa, data related to illness awareness and other clinical, cognitive and psychosocial variables will be collected longitudinally in the 3 and 6 months after.

Finally, a quantitative analysis of the results obtained will be carried out.

DETAILED DESCRIPTION:
Lack of illness awareness in patients suffering from eating disorders is a recognized phenomenon that has received abundant theoretical interest in recent decades. However, research on the subject is limited and has provided inconsistent results.

Illness denial rates reported in different studies have yielded discrepant figures ranging from 15% to 80% in anorexia nervosa. Attempts have been made to explain this variability between results by the use of dichotomous classifications and inconsistent or unspecified criteria to designate patients as deniers or admitters. Some authors suggest higher rates of impaired insight in eating disorders, assuming greater impairment in people who refuse or do not demand treatment and who were not included in these studies.

Moreover, the relationship between the lack of insight, the evolution of the disorder and the fluctuations of other clinical variables, such as affective symptomatology or body mass índex, cognitive and psychosocial variables, has not been clearly established. In a recent cross-sectional study, no relationship was found between insight and the duration of the disease in patients with anorexia nervosa, suggesting that there could be deterioration in both early and chronic phases.

To date, only two longitudinal studies have been conducted on insight in eating disorders. According to these studies, the variation in illness awareness remains relatively stable over time, but despite this, its relationship with changes in nutritional status is not clear.

Regarding the development of specific tools to assess insight in eating disorders, there is only one recently created scale in English, the Schedule for the Assessment of Insight in Eating Disorders (SAI-ED), by Konstantakopoulos (2020). This scale was initially created as an adaptation of the SAI-E for psychosis, it includes 8 items to be assessed by a clinician, easy to apply as it does not require prior training and it has been shown to have good psychometric properties. To date, no adaptation's study of this scale for the Spanish population was conducted.

Objective: To study the characteristics of illness awareness, its dimensions and its evolution in relation to clinical, cognitive and psychosocial variables in patients with anorexia nervosa.

Design: observational longitudinal design. Method: First, the process of translating and culturally adapting the SAI-ED scale to Spanish will be carried out and, over 9 months, patients who are admitted to the Eating Disorders Unit of the Hospital de la Santa Creu i Sant Pau (HSCSP) and the Eating Disorders Unit of the H. Mutua de Terrassa will be offered to participate in the study. Through individual clinical interviews and self-reports, a first sample will be collected to allow the validation study of the scale in the Spanish population.

The sample will include patients with Anorexia Nervosa and Bulimia Nervosa who understand and speak Spanish or Catalan and sign the informed consent for participation. Participants will be recruited consecutively until N=80 is reached.

From a subsample of patients with anorexia nervosa, data related to illness awareness and other clinical, cognitive and psychosocial variables will be collected longitudinally in the 3 and 6 months after.

Finally, a quantitative analysis of the results obtained will be carried out.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of bulimia nervosa, anorexia nervosa or atypical anorexia nervosa according to Diagnostic and Statistical Manual (DSM-5) criteria.
* Age between 18 and 65 years.
* Female sex.

Exclusion Criteria:

* Comorbid neurological disorder.
* Clinical worsening requiring hospitalization.
* Patients who do not give consent.
* Patients who do not understand or speak Spanish or Catalan.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The subjects of the initial cross-sectional study will be patients with anorexia or bulimia recruited consecutively from the Eating Disorder Unit of the Hospital de la Santa Creu i Sant Pau (HSCSP) and from the Hospital Universitari Mútua de Terrassa (HUMT). A sub-sample of the study patients diagnosed with anorexia or atypical anorexia will participate in the longitudinal follow-up.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Insight impairment | Baseline and 6 months.
  Change from Baseline Illness awareness impairment in patients with an eating disorder measured at 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided